CLINICAL TRIAL: NCT01812967
Title: Mechanism of Action of Milk and Its Components on Glycemic Control in Healthy Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Purpose: Prevention
Other Study IDs: Milk Components Study
Record Dates: First submitted 2013-03-13; First posted 2013-03-18 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Glycemic Control; Gastrointestinal Hormone Response; Healthy Young Men
MeSH Terms: interventions — Milk Proteins; Lactose

INTERVENTIONS:
Dietary Supplement: Milk Fat
Dietary Supplement: Milk Protein
Dietary Supplement: Lactose
Other: Whole milk (3.25% M.F.( — Commercially available milk from the grocery store
Dietary Supplement: Simulated Milk Beverage — Added lactose + fat + protein together to form a mixture

SUMMARY:
The investigators hypothesize that the physiological effects of milk on satiety and glycemic control are mediated by the interaction between its macronutrient components by both insulin-dependent and independent mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young men
* 20-30 years of age
* BMI: 20-24.9 kg/m2

Exclusion Criteria:

* Smoking
* Dieting
* Skipping breakfast
* Lactose intolerance or allergies to milk
* Taking medications that may affect glucose metabolism or appetite
* Diabetes (fasting blood glucose ≥ 7.0 mmol/L) or other metabolic diseases

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Glucose | 0-180 min

SECONDARY OUTCOMES:
Insulin | 0-180 min

OTHER OUTCOMES:
Gastrointestinal hormones and gastric emptying rate | 0-180 min
  Gatrointestinal hormones measured include plasma concentrations of glucagon-like peptide-1 (GLP-1), peptide tyrosine tyrosine (PYY), cholecystokinin (CCK), and ghrelin.
  Gastric emptying is assessed indirectly by adding 1.5 g of paracetamol (acetaminophen) to each beverage and measuring plasma paracetamol concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Panahi S, El Khoury D, Kubant R, Akhavan T, Luhovyy BL, Goff HD, Anderson GH. Mechanism of action of whole milk and its components on glycemic control in healthy young men. J Nutr Biochem. 2014 Nov;25(11):1124-1131. doi: 10.1016/j.jnutbio.2014.07.002. Epub 2014 Jul 31. PMID 25167977